CLINICAL TRIAL: NCT00065793
Title: VLDL and LDL Particle Types as Coronary Heart Disease Risk Factors
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank M. Sacks, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1232; R01HL070159 (NIH)
Record Dates: First submitted 2003-07-31; First posted 2003-08-04 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Diabetes Mellitus; Diabetes Mellitus, Non-insulin Dependent
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To evaluate very low density lipoprotein (VLDL) and low density lipoprotein (LDL) particle types as predictors of initial coronary events.

DETAILED DESCRIPTION:
BACKGROUND:

Plasma triglyceride concentration is an independent although relatively weak risk factor for coronary heart disease (CHD). The relative weakness of plasma triglycerides to predict CHD may be due to the substantial diversity of lipoprotein particles that carry the triglycerides, some being related to atherosclerosis and CHD more than others. The investigators have shown in patients who have had a myocardial infarction that the rather weak association between triglycerides and subsequent coronary events is secondary to a stronger relationship with specific types of VLDL remnants, those in the LDL density range that contain apoCIIl.

DESIGN NARRATIVE:

The study will evaluate VLDL and LDL particle types as predictors of initial coronary events in men from the Health Professional Follow-up Study (HPFS) and women from the Nurses Health Study (NHS). A prospective nested case-control design will be used with a total of 1000 CHD cases and 1000 matched controls, with equal numbers of men and women. The investigators will specifically investigate the role of apoCIII containing VLDL and LDL particles in diabetes by over sampling so that 50% of the patients will have type 2 diabetes mellitus. Their previous work shows that LDL apoCIII particles are independent predictors of recurrent CHD in diabetic patients who survived a myocardial infarction. They hypothesize that apoCIII may have a special role in dyslipidemia and CHD in diabetes. Secondary Aims: Besides apoCIII, other small apolipoproteins, apo C1, CII, and All are components of VLDL and LDL and modulate the metabolism of apoB lipoproteins. It is likely that these apolipoproteins have a relationship with human atherosclerosis. They will measure these apolipoproteins in VLDL and LDL and evaluate their relationship to CHD. They will also investigate the associations between these new lipoprotein risk factors and intake of foods and nutrients, physical activity, and other risk factors, including smoking, BMI, age and gender. The results will provide new means to identify nondiabetic and diabetic persons who are at high risk of developing CHD and the environmental determinants, and could form the basis for new lipoprotein targets for lipid management by diet and medicines.

ELIGIBILITY:
Cases having first coronary event

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses Health Study Health Professionals Follow-up Study
Sampling Method: Non-Probability Sample
Enrollment: 1478 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
apoB concentration of LDL with apoC-III | 10-14 years
  observational follow-up for coronary events

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sacks, MD, Principal Investigator — Harvard School of Public Health (HSPH); Frank Sacks, MD, Principal Investigator — Brigham and Women's Hospital